CLINICAL TRIAL: NCT04648449
Title: Artificial Intelligence (AI) Support in Medical Emergency Calls - "The AISMEC-study" -Can Artificial Intelligence Improve the Precision in Identifying Acute Stroke in Emergency Medical Calls?
Brief Title: Artificial Intelligence (AI) Support in Medical Emergency Calls
Acronym: AISMEC
Status: Active, not recruiting | Type: Observational
Sponsor: Haukeland University Hospital (Other)
Collaborators: Helse Vest (Other); Western Norway University of Applied Sciences (Other); Oslo University Hospital (Other); The Norwegian Heart and Lung Patient Organization (Unknown); Helsetjenestens driftsorganisasjon for nødnett HF (HDO) (Unknown); The Norwegian Stroke Register (Unknown)
Responsible Party: Sponsor
Other Study IDs: 108573
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-03

CONDITIONS: Stroke, Acute; Apoplexy; Brain; Emergencies; Communication, Multidisciplinary
Keywords: EMCC; Stroke; Apoplexy; Emergency Medical Service Communication Systems; Dispatch; Artificial intelligence; Machine learning
MeSH Terms: conditions — Stroke; Emergencies; Communication

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Artificial intelligence on emergency calls — AI listens to all calls to Bergen EMCC, detecting calls regarding possible stroke.

SUMMARY:
More than 12.000 patients suffer acute stroke in Norway every year, but less than half of them reach hospital within the current treatment window for thrombolysis. Stroke is the third-highest cause of death and the number one cause of severe disability requiring long time care at institutions. Consequently this has a high impact on society, patients and relatives, in addition to high costs related to care estimated to approximately 10 billion NOK per year. Although there are few studies on emergency medical communication centres (EMCC) in Norway, some have shown that the performance of the emergency medical communication centres can be improved. This project will seek to amend EMCC´s handling of acute stroke inquiries using artificial intelligence (AI), thus contributing to getting the patient to hospital in time for optimal treatments.

DETAILED DESCRIPTION:
In this project, the investigators will collect data from all stroke patients discharged from Helse Bergen in 2019 (approx. 1000 patients) via the Norwegian Stroke Registry (NSR). For these patients, structured hospital data from Helse Bergen will be retrieved, and based on these and the spoken content of their emergency call regarding the stroke, the investigators will use machine learning to calculate the stroke risk. The connection of historical hospital data to the spoken words in the emergency call, amplifies the analysis of emergency calls in a novel way, in comparison to sound analysis alone.

After retrieving and connecting stroke patient data, the investigators train the deep network using data from 2019. Accordingly, testing will be performed based on patients from the first half of 2020. A separation of the data into training, test, and validation assures that our trained network does not over fit on the training data and can reproduce similar results on previously unseen patients. Finally, the investigators will compare the performance of the AI with the current system through statistical analyses on data from a period of approximately one year of live usage of the AI in AMK Bergen. This will enable us to evaluate to what degree the system is able to improve within the decision process of the EMCC operators in terms of sensitivity and specificity.

Summarized, the primary objective is to build a robust, working prototype of an AI system capable of real-time identification of acute stroke for improved assessment in emergency medical calls.

Our secondary objectives are:

* To implement an AI system capable of providing fast prediction of whether a patient is suffering from acute stroke or not based on audio from emergency call and available data sources within the hospital records
* To prove that AI systems can be used to assist and improve the triage decision procedure of the EMCC operator.

The anticipated result is to deliver fast (i.e. seconds) prediction scores to assist the EMCC operator in recognizing acute stroke patients, which provides an improved sensitivity and specificity compared to manual assessment only.

ELIGIBILITY:
Inclusion Criteria:

* All callers to medical emergency number 113 in Bergen

Exclusion Criteria:

* Age <18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All calls to 113 in Bergen will be subject to the AI. A warning will be given the EMCC-operator if risk of stroke, when combining contents in the call and historical data in the hospital record, exceeds a certain limit.
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Stroke recognition in medical emergency calls | Sept. 22 - Sept. 23
  Survey AI's ability to recognize stroke, compared to the current system

CONTACTS AND LOCATIONS:
Overall Officials: Guttorm Brattebo, Professor II, Study Director — Haukeland University Hospital
Locations (1):
- Haukeland Universitetssykehus, Kirurgisk serviceklinikk, Nasjonalt kompetansesenter for helsetjenestens kommunikasjonsberedskap, Bergen, Bergen, Norway

IPD SHARING:
Plan to Share IPD: No
Not relevant at this stage.